CLINICAL TRIAL: NCT07358676
Title: An Exploratory Phase II Study of Bemotuzumab Combined With Chemotherapy and Anlotinib as Induction Therapy, Followed by Bemotuzumab, Anlotinib, and Consolidative Thoracic Radiotherapy in Patients With Extensive-Stage Small Cell Lung Cancer
Brief Title: A Study of Bemotuzumab Plus Chemotherapy and Anlotinib Induction Followed by Bemotuzumab, Anlotinib and Consolidative Thoracic Radiotherapy in Extensive-Stage Small Cell Lung Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E20260033
Record Dates: First submitted 2026-01-14; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Small Cell Lung Cancer (SCLC); SCLC, Extensive Stage
Keywords: Small Cell Lung Cancer (SCLC); bemotuzumab; anlotinib; hypofractionated radiotherapy; Induction therapy
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — anlotinib; Drug Therapy; Radiotherapy; Radiation Dose Hypofractionation

STUDY DESIGN:
Intervention Model Description: This is a single-arm, exploratory study. All enrolled participants receive the same intervention sequence.
Masking Description: This is an open-label study. No masking (blinding) is used.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental Group (Experimental): Participants receive a multi-phase experimental regimen. Induction (4 cycles, q3w): Bemotuzumab (1200 mg IV, Day 1) combined with investigator's choice of platinum-etoposide chemotherapy (Carboplatin AUC=5 or Cisplatin 75-80 mg/m² on Day 1, plus Etoposide 100 mg/m² IV on Days 1-3) and oral Anlotinib (12 mg once daily on Days 1-14, then 7 days off).
  Consolidation (2 cycles, q3w): Bemotuzumab (same dose) + Anlotinib (same schedule) with concurrent hypofractionated thoracic radiotherapy (5 Gy per fraction for 5 fractions).
  Maintenance: Bemotuzumab (q3w) + Anlotinib (same schedule) until disease progression, unacceptable toxicity, or other withdrawal criteria. Anlotinib dose may be reduced (12mg → 10mg → 8mg) for managing toxicity.
  Interventions: Combination Product: Bemotuzumab + Anlotinib + Chemotherapy + Radiotherapy

INTERVENTIONS:
Combination Product: Bemotuzumab + Anlotinib + Chemotherapy + Radiotherapy — This is a multi-phase combined modality regimen.
  Induction Phase (4 cycles): Bemotuzumab (1200mg IV, Day1 q3w) + Platinum/Etoposide chemotherapy (Carboplatin [AUC5] or Cisplatin [75-80 mg/m²] on Day1, plus Etoposide [100 mg/m² IV, Days1-3]) + oral Anlotinib (12mg, Days1-14, then 7 days off).
  Consolidation Phase (2 cycles): Bemotuzumab (same dose) + Anlotinib (same schedule) + concurrent Thoracic Radiotherapy (5 Gy per fraction for 5 fractions).
  Maintenance Phase: Bemotuzumab (q3w) + Anlotinib until disease progression or unacceptable toxicity.
  Anlotinib Dose Modification: The dose may be increased to 12mg if well tolerated. For toxicity, it can be reduced sequentially (12mg→10mg→8mg). Treatment is discontinued if 8mg is not tolerated. For subjects at 8mg, one dose re-escalation is permitted if, in the investigator's judgement, clinical benefit is possible and safety is stable.
  Other Names: Anlotinib Hydrochloride; Bemotuzumab Injection; Fucovee; Hypofractionated Radiotherapy

SUMMARY:
This is a phase II study evaluating a new combination therapy for untreated extensive-stage small cell lung cancer. The treatment involves an initial phase with the drug Bemotuzumab plus standard chemotherapy and anlotinib, followed by a phase combining Bemotuzumab, anlotinib, and chest radiation. The primary objectives are to assess the efficacy of this approach in delaying cancer growth (progression-free survival) and to evaluate its safety in approximately 25 patients.

DETAILED DESCRIPTION:
This is an exploratory Phase II clinical trial for previously untreated extensive-stage small cell lung cancer (ES-SCLC). The study evaluates a novel three-phase sequential treatment strategy: patients first receive induction therapy with Bemotuzumab combined with standard chemotherapy and Anlotinib; those achieving disease control then proceed to consolidation therapy with Bemotuzumab, Anlotinib, and concurrent thoracic radiotherapy; followed by a maintenance phase with Bemotuzumab plus Anlotinib. The primary objectives are to assess the regimen's efficacy in prolonging progression-free survival (PFS) and to observe its safety profile. The study plans to enroll approximately 25 patients.

ELIGIBILITY:
**Inclusion Criteria:**

1. Histologically or cytologically confirmed extensive-stage small cell lung cancer (ES-SCLC) per VALG staging.
2. No prior systemic therapy for ES-SCLC.
3. At least one measurable lesion as defined by RECIST 1.1 criteria.
4. Age 18-75 years.
5. ECOG performance status of 0-2.
6. Life expectancy of ≥3 months.
7. Adequate hematologic and organ function:

   * Absolute neutrophil count (ANC) ≥ 1.5 × 10^9/L.
   * Platelet count ≥ 100 × 10^9/L.
   * Hemoglobin ≥ 80 g/L.
   * Creatinine clearance ≥ 50 mL/min.
   * Total bilirubin ≤ 1.5 × upper limit of normal (ULN).
   * AST and ALT ≤ 2.5 × ULN.
   * Albumin ≥ 28 g/L.
   * INR and APTT ≤ 1.5 × ULN.
   * Left ventricular ejection fraction (LVEF) ≥ 50%.
8. For females of childbearing potential: negative serum pregnancy test within 3 days prior to dosing and agreement to use highly effective contraception.
9. For males: agreement to use barrier contraception.
10. Willing and able to provide written informed consent and comply with study procedures.

**Exclusion Criteria:**

1. Symptomatic brain metastases. (Asymptomatic, treated, and stable brain metastases for ≥1 month without steroids are allowed).
2. Prior thoracic radiotherapy for SCLC.
3. Prior treatment with anti-angiogenic agents (e.g., anlotinib, bevacizumab) or anti-PD-1/PD-L1 therapies.
4. Factors affecting oral medication intake (e.g., inability to swallow, major gastrointestinal resection).
5. Uncontrolled effusions requiring repeated drainage (pleural, pericardial, or ascites).
6. Imaging evidence of tumor invasion of major blood vessels or high risk of fatal hemorrhage as judged by the investigator.
7. History of significant bleeding tendency or coagulopathy, including clinically significant hemoptysis (>1 tablespoon daily within 3 months) or significant bleeding within 4 weeks prior to enrollment.
8. Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to enrollment.
9. Arterial/venous thrombotic events within 6 months prior to enrollment (e.g., cerebrovascular accident, deep vein thrombosis, pulmonary embolism).
10. Active autoimmune disease requiring systemic treatment within 2 years prior to first dose.
11. Any other condition that, in the investigator's judgment, increases risk or renders the patient unsuitable for the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2027-01-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) | From enrollment until disease progression or death from any cause, assessed up to approximately 24 months.
  PFS is defined as the time from enrollment to the first documented disease progression according to RECIST 1.1 criteria or death from any cause, whichever occurs first. Tumor assessments are performed every 6 weeks (every 2 treatment cycles).

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | From enrollment until the first documented CR or PR, assessed up to approximately 24 months.
  ORR is defined as the proportion of participants who achieve a best overall response of Complete Response (CR) or Partial Response (PR) as assessed by the investigator according to RECIST 1.1 criteria.
Overall Survival (OS) | From enrollment until death from any cause, assessed up to approximately 24 months.
  OS is defined as the time from enrollment to death from any cause.
Incidence of Grade ≥3 Immune-Related Adverse Events (irAEs) | From first dose of study drug until 28 days after the last dose, assessed up to approximately 24 months.
  The incidence of treatment-emergent adverse events assessed as immune-related and graded ≥3 according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Dingzhi Huang, Doctor, Principal Investigator — Tianjin Medical University Cancer Institute and Hospital; Ningbo Liu, Doctor, Principal Investigator — Tianjin Medical University Cancer Institute and Hospital
Locations (1):
- Tianjin Medical University Cancer Institute & Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data for all primary and secondary outcome measures will be made available.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be available within 6 months of study completion
Access Criteria: Data access requests will be reviewed by an external independent review panel. Requestors will be required to sign a Data Access Agreement.